CLINICAL TRIAL: NCT03968692
Title: Study of the Adequacy of the Requests of Prostate-Specific Antigen (PSA), Factors Associated With the False Negative and Positive Results and the Impact on Patient's Health
Brief Title: Adequacy of Prostate-Specific Antigen (PSA) Requests
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Hospital Universitario San Juan de Alicante (Other); Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Blanca Juana Lumbreras Lacarra, Professor of Preventive Medicine and Public Health, Universidad Miguel Hernandez de Elche
Other Study IDs: PI17/01883.1; PI17/01883 (Other Grant/Funding Number: MINECO-FEDER)
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Prostate-Specific Antigen
Keywords: Prostatic Neoplasms; Practice Guideline; Early Detection of Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Diagnostic Test: Prostate-Specific Antigen test — Prostate-Specific Antigen (PSA) test as opportunistic screening or in the presence of symptoms

SUMMARY:
Objectives.

The primary aim of this study is to evaluate the characteristics of the determination of PSA for the early detection of prostate cancer or in the presence of symptoms, in general practice in two health departments of the Valencian Community (Spain).

Specific objectives:

* To describe the PSA determinations that are performed in clinical practice, with the exception of patients with prostate cancer or who are being followed for previous high PSA values.
* To study the adequacy of PSA requests according to the available recommendations, considering sociodemographic and clinical aspects of the patient, such as the time interval since the last PSA test.

The investigators will randomly select patients from the Health Departments 17 and 19, in the Valencian Community (Spain) with a PSA request from Primary health centres.

DETAILED DESCRIPTION:
Sample size and recruitment procedure:

During the last semester of 2016, 9,963 PSA determinations were carried out at Sant Joan d'Alacant Hospital and a similar number at Alicante General Hospital. Primary health centres requested most determinations. The prevalence of prostate cancer in 2012 was 527.3/100,000 men in Spain. Considering that there are about 120,000 men in each of the included Departments of Health, approximately 630 men will have the diagnosis of prostate cancer in each of them.

According to the established recommendations, a patient with prostate cancer had a PSA determination every 3-6 months. Consequently, 1,260 determinations per centre would correspond to prostate cancer patients each 6 months. Therefore, the investigators would have in each department approximately 8,740 determinations of patients without prostate cancer, and therefore, possible candidates to enter in our study.

According to a pilot study with 360 patients in which 35.6% of the requested PSA determinations do not follow the available recommendations with a 95% margin of error and 2% accuracy, the investigators will include a total of 1,410 determinations from the two centres. Hence, for the determination of specific objective 1, the investigators will select a random sample of 705 patients with a PSA determination in each centre.

From each clinical analysis laboratory, the investigators will randomly select 300 primary care analyses with PSA determination for each month from January to April 2018. The investigators will select the patients who satisfy the inclusion criteria consecutively from this list until 180 are included.

Data collection procedure:

The investigators will collect the following variables from the medical records for each patient: Demographic characteristics, setting (primary care or clinical service), PSA tests carried out in the last 12 months and PSA value, anthropometric measures and other comorbidities.

The investigators will analyze the appropriateness of PSA determinations according to the criteria established by the clinical practice guidelines of the EAU, and the May 2018 update of the USPSTF. All the reviewers are trained in the use of these guidelines.

A pilot study of a sample of 30 determinations will be independently evaluated by the nine researchers the application of the determined criteria. If the agreement is high, the rest of the determinations will be evaluated separately by at least two researchers using a predesigned google form. In case of disagreement between two of the evaluators, the case will review by a third, or discussed in a joint meeting with the rest of the team.

Data analysis plan:

The analysis will be performed using the Stata IC 15 program. The investigators will estimate the frequency and 95% confidence interval of the adequacy of PSA determinations to established recommendations. The investigators will evaluate the inter-observer agreement in the determination of adequacy using the Kappa index. In order to assess the relationship with potential explanatory variables, and the magnitude of the association, the investigators will calculate prevalence ratios. If necessary, a log-binomial regression will be performed to get an adjusted analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a PSA determination requested in a routine health examination from primary health centers from the Health Department 17 and 19, in the Valencian Community (Spain).

Exclusion Criteria:

* Patients who have been previously diagnosed with prostate cancer.
* Patients who are being followed for previous high PSA values.

Ages: 18 Years to 99 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Men over 18 from the Health Department 17 and 19, in the Valencian Community (these include General University Hospital of Sant Joan d'Alacant and General University Hospital of Alicante, respectively). These are referral hospitals for all individuals living in their catchment areas and belong to the National Health Care System (the majority of the population in Spain uses the National Health System (NHS) as the main medical service (the publicly funded insurance scheme covers 98.5% of the Spanish population).
  We have not established maximum age limit.
Sampling Method: Probability Sample
Enrollment: 1410 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Appropriateness of PSA determinations according to the criteria established by the clinical practice guidelines of the EAU, and the May 2018 update of the USPSTF | 6 months
  We define appropriateness of the PSA determination as follows:
  1. Presence of symptoms suggestive of prostate pathology (difficulty starting to urinate; weak or interrupted urine flow; frequent urination, especially at night; difficulty emptying the bladder completely; pain or burning when urinating; blood in the urine or semen; persistent pain in the back, hips, or pelvis; pain when ejaculating, and erectile dysfunction);
  2. Patients in opportunistic screening defined by satisfaction of the criteria of at least one of the two guidelines:
     1. Age 55-69 years (USPSTF) or older than 50 years and a life expectancy of at least 10 years, provided that have not had a PSA determination in the last 24 months (EAU).
     2. Patients under 55 years of age (USPSTF) or patients from 45 to 50 years old with a family history of first degree and/or African American race, provided that have not had a PSA determination in the last 24 months (EAU).

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - San Juan de Alicante Hospital, Sant Joan d'Alacant, Alicante
  - FISABIO, Alicante

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ren JS, Masuyer E, Ferlay J. Global estimates of cancer prevalence for 27 sites in the adult population in 2008. Int J Cancer. 2013 Mar 1;132(5):1133-45. doi: 10.1002/ijc.27711. Epub 2012 Jul 26. PMID 22752881